CLINICAL TRIAL: NCT01956591
Title: Retrospective Evaluation of Long Term Use of Oxybutynin in the Pharmacological Treatment of Primary Hyperhidrosis
Brief Title: Long Term Results of the Use of Oxybutynin for the Treatment of Hyperhidrosis
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Nelson Wolosker, PhD, Hospital Israelita Albert Einstein
Other Study IDs: HIsraelitaAE
Record Dates: First submitted 2013-08-16; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Hyperhidrosis
Keywords: Treatment efficacy; Long-term effects; Tachyphylaxis; Undesirable effects; Side effects; Self-assessment; Hyperhidrosis; Quality of life
MeSH Terms: conditions — Hyperhidrosis | interventions — oxybutynin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Axillary hyperhidrosis: Patients whose major complaint is excessive sweating in the axillary region (i.e, sweating in the armpit). Patients that also have hyperhidrosis - but that are less bothersome on other sites (e.g., palmar hyperhidrosis) are not excluded, but are accounted for accordingly to their main complaint.
  Interventions: Drug: Oxybutynin
- Palmar hyperhidrosis: Patients whose major complaint is excessive sweating in the palmar region (i.e, sweating in the hands). Patients that also have hyperhidrosis - but that are less bothersome on other sites (e.g., axillary hyperhidrosis) are not excluded, but are accounted for accordingly to their main complaint.
  Interventions: Drug: Oxybutynin
- Plantar hyperhidrosis: Patients whose major complaint is excessive sweating in the plantar region (i.e, sweating in the feet). Patients that also have hyperhidrosis - but that are less bothersome on other sites (e.g., axillary hyperhidrosis) are not excluded, but are accounted for accordingly to their main complaint.
  Interventions: Drug: Oxybutynin
- Cranio-facial hyperhidrosis: Patients whose major complaint is excessive sweating in the cranio-facial region (i.e, sweating in the face). Patients that also have hyperhidrosis - but that are less bothersome on other sites (e.g., axillary hyperhidrosis) are not excluded, but are accounted for accordingly to their main complaint.
  Interventions: Drug: Oxybutynin
- Other sites hyperhidrosis: Patients whose major complaint is excessive sweating in other sites of the body (e.g., on the chest, on the abdomen). Patients that also have hyperhidrosis - but that are less bothersome on other sites previously grouped (e.g., axillary hyperhidrosis) are not excluded, but are accounted for accordingly to their main complaint.
  Interventions: Drug: Oxybutynin

INTERVENTIONS:
Drug: Oxybutynin — All patients are treated with oxybutynin for hyperhidrosis. Usual maintenance dose is 10mg/day, but dose may vary according to weight, efficacy and side effects. Our standard protocol starts with 2.5mg/day in the first 7 days, progresses to 5mg/day for 14 days and then reaches the usual maintenance dose of 10mg/day afterwards.

SUMMARY:
Evaluate the long term efficacy and side effects of oxybutynin in the treatment of hyperhidrosis.

DETAILED DESCRIPTION:
This retrospective study aims to evaluate the medical charts of patients who were treated with oxybutynin for at least six months for primary hyperhidrosis. The investigators variables of interest are: (1) quality of life before pharmacological therapy and after six weeks, (2)self-perception of improvement in hyperhidrosis after six weeks of treatment and on last visit (whenever this occur, as long as this happens after six months), (3) side effects related to drug use.

ELIGIBILITY:
Inclusion Criteria:

* Primary hyperhidrosis
* At least 180 days of treatment with oxybutynin

Exclusion Criteria:

* Incomplete medical chart
* Patients with glaucoma

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Out-patients on two tertiary hospitals (Hospital Israelita Albert Einstein and Hospital das Clínicas - HCFMUSP) who seeked medical attention because of hyperhidrosis.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2007-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Quality of life | 1 day before treatment
  Evaluate the Quality of life (using a standardized questionnaire for hyperhidrotic patients) before pharmacological treatment
Quality of life | Forty-two days after treatment
  Evaluate the Quality of life (using a standardized questionnaire for hyperhidrotic patients) after 42 days of treatment

SECONDARY OUTCOMES:
Perception of improvement in excessive sweating | After 42 days of treatment
  We want to analyze the patient's self perception (grades 0 to 10) of amelioration in sweating after forty-two days of treatment
Perception of improvement in excessive sweating | 1 day (On the last medical visit)
  We want to analyze the patient's self perception (grades 0 to 10) of amelioration in sweating on the last medical visit (whenever this happens).

OTHER OUTCOMES:
Side effects in the use of oxybutynin for hyperhidrosis | After 42 days of treatment
  Assess the side effects that have been reported on patient's charts, such as: dry mouth, constipation, headache, glaucoma, bowel obstruction and any other side effect reported
Side effects in the use of oxybutynin for hyperhidrosis | 1 day )On the last medical visit)
  Assess the side effects that have been reported on patient's charts, such as: dry mouth, constipation, headache, glaucoma, bowel obstruction and any other side effect reported on the last medical return of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Wolosker, PhD, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Wolosker N, Schvartsman C, Krutman M, Campbell TP, Kauffman P, de Campos JR, Puech-Leao P. Efficacy and quality of life outcomes of oxybutynin for treating palmar hyperhidrosis in children younger than 14 years old. Pediatr Dermatol. 2014 Jan-Feb;31(1):48-53. doi: 10.1111/pde.12142. Epub 2013 Apr 29. PMID 23627681
- [Background] Wolosker N, de Campos JR, Kauffman P, Yazbek G, Neves S, Puech-Leao P. Use of oxybutynin for treating plantar hyperhidrosis. Int J Dermatol. 2013 May;52(5):620-3. doi: 10.1111/j.1365-4632.2012.05746.x. PMID 23590378
- [Background] Wolosker N, Krutman M, Campdell TP, Kauffman P, Campos JR, Puech-Leao P. Oxybutynin treatment for hyperhidrosis: a comparative analysis between genders. Einstein (Sao Paulo). 2012 Oct-Dec;10(4):405-8. doi: 10.1590/s1679-45082012000400002. English, Portuguese. PMID 23386077
- [Background] Wolosker N, de Campos JR, Kauffman P, Puech-Leao P. A randomized placebo-controlled trial of oxybutynin for the initial treatment of palmar and axillary hyperhidrosis. J Vasc Surg. 2012 Jun;55(6):1696-700. doi: 10.1016/j.jvs.2011.12.039. Epub 2012 Feb 16. PMID 22341836
- [Background] Wolosker N, de Campos JR, Kauffman P, Neves S, Munia MA, BiscegliJatene F, Puech-Leao P. The use of oxybutynin for treating axillary hyperhidrosis. Ann Vasc Surg. 2011 Nov;25(8):1057-62. doi: 10.1016/j.avsg.2011.06.007. PMID 22023940
- [Background] Wolosker N, Campos JR, Kauffman P, Munia MA, Neves S, Jatene FB, Puech-Leao P. The use of oxybutynin for treating facial hyperhidrosis. An Bras Dermatol. 2011 May-Jun;86(3):451-6. doi: 10.1590/s0365-05962011000300005. PMID 21738960
- [Background] Wolosker N, de Campos JR, Kauffman P, Neves S, Yazbek G, Jatene FB, Puech-Leao P. An alternative to treat palmar hyperhidrosis: use of oxybutynin. Clin Auton Res. 2011 Dec;21(6):389-93. doi: 10.1007/s10286-011-0128-4. Epub 2011 Jun 19. PMID 21688168
- [Background] Try C, Messikh R, Elkhyat A, Aubin F, Humbert RP. [Use of oral oxybutynin at 7.5 mg per day in primary hyperhidrosis]. Rev Med Liege. 2012 Oct;67(10):520-6. French. PMID 23167161
- [Background] Maillard H, Fenot M, Bara C, Celerier P. [Therapeutic value of moderate-dose oxybutynin in extensive hyperhidrosis]. Ann Dermatol Venereol. 2011 Oct;138(10):652-6. doi: 10.1016/j.annder.2011.07.002. Epub 2011 Aug 17. French. PMID 21978500
- [Background] Lefrandt JD, Maurer JM. Oxybutynin for hyperhidrosis. Neth J Med. 2007 Oct;65(9):356. No abstract available. PMID 17954957
- [Background] Schollhammer M, Misery L. Treatment of hyperhidrosis with oxybutynin. Arch Dermatol. 2007 Apr;143(4):544-5. doi: 10.1001/archderm.143.4.544. No abstract available. PMID 17438194
- [Background] Mijnhout GS, Kloosterman H, Simsek S, Strack van Schijndel RJ, Netelenbos JC. Oxybutynin: dry days for patients with hyperhidrosis. Neth J Med. 2006 Oct;64(9):326-8. PMID 17057269
- [Background] Tupker RA, Harmsze AM, Deneer VH. Oxybutynin therapy for generalized hyperhidrosis. Arch Dermatol. 2006 Aug;142(8):1065-6. doi: 10.1001/archderm.142.8.1065. No abstract available. PMID 16924061